CLINICAL TRIAL: NCT03431870
Title: Prospective Study to Examine the Impact of Anesthesia on the Dimension of the Ascending Aorta in Patients With a Dilated Aorta Who Undergo Open-heart Surgery
Brief Title: Impact of Anesthesia on the Dimension of the Ascending Aorta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-18-4459-ER-CTIL
Record Dates: First submitted 2018-01-23; First posted 2018-02-13 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aorta dilated (Other): Patients with aorta of 40mm or more who undergo a cardiac surgery. The intervention include: Trans-Esophageal Echocardiography
  Interventions: Other: Trans-esophageal echocardiography

INTERVENTIONS:
Other: Trans-esophageal echocardiography — Perform a trans-esophageal echocardiography before and after anesthesia.
  Other Names: Cardiac surgery

SUMMARY:
The aim of this study is to evaluate the accuracy and reliability of intra-operative TEE after the induction of anesthesia when assessing proximal thoracic aorta diameters in a cohort of aortic aneurysm patients.

DETAILED DESCRIPTION:
Dilatation of the ascending aorta often progresses silently in an asymptomatic patient, until an acute complication occurs (such as a dissection or rupture), which is directly related to the diameter of the aortic. To prevent these extremely harmful situations, aortic replacement surgery, as indicated by significant dilatation of the ascending aorta, could be the option of choice (1). The decision to perform elective surgery depends on the measurement of the thoracic aorta diameter, which would rely on the largest aortic dimension. Trans-thoracic echocardiography (TTE) is widely used to assess the aortic root (2), and results from computed tomography (CT) scans are used to evaluate the ascending aorta beyond the sinotubular junction (3, 4). Both these tests facilitate follow-up evaluation of patients with thoracic aortic aneurysm. Usually, patients are referred for surgery based on the findings of one or both of these examinations. Furthermore, when a patient is referred for surgery, intra-operative trans-esophageal echocardiography (TEE) is often performed after induction of the anesthesia in order to evaluate the aortic dimension and valve function.

In some cases, the diameter of the aorta is considered borderline for replacement, in which case the TEE measurement could reverse the decision-making, especially when the indication for surgery is due to valve pathology, with the aorta being a secondary consideration.

From the investigators experience, intra-operative TEE aortic measurements after the anesthesia are not entirely accurate, and could under-estimate the diameter of the aorta. Relying on intra-operative TEE measurements could result in under-treatment of the dilated aorta, especially when its replacement is secondary to other cardiac pathologies (e.g. AVR, CABG) that require surgery.

Influence of intra-operative anesthesia on TEE measurements of the aorta are not described in the current literature. If the investigators hypothesis is correct, adjustments will need to be made regarding the surgical management of patients with borderline aortic dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Ascending aorta of 40 mm and above
* Patients who undergo cardiac surgery

Exclusion Criteria:

* Unstable patients
* Patients who underwent a previous cardiac surgery
* Patients who were diagnosed with aortic dissection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2022-01-21 (Estimated); Study Completion 2022-01-21 (Estimated)

PRIMARY OUTCOMES:
difference in the aortic dimension | intraoperative
  10% difference in the aortic dimension before and after anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Eilon Ram, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No